CLINICAL TRIAL: NCT05178953
Title: The Therapeutic Effect of Co-administration of Pentoxifylline and Zinc on Semen Parameters, Reproductive Hormones, DNA Fragmentation, and Some Biochemical, and Inflammatory Parameters in Men With Idiopathic Infertility
Brief Title: The Therapeutic Effect of Co-administration of Pentoxifylline and Zinc in Men With Idiopathic Asthenozoospermia
Acronym: PTX-Zn
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arak University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zeynab, Principal Investigator, Arak University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1898
Record Dates: First submitted 2021-12-15; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Men Infertility
MeSH Terms: interventions — Zinc Sulfate; Zinc; Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pentoxifylline group (Experimental): Group 1: Patients receiving pentoxifylline (TRENTAL 400 mg tablets, OSPS; 400 mg, twice daily) Infertile men referred to an infertility treatment center who have had unprotected sex for at least one year have not had normal fertility in their partner. These men are all married. According to WHO criteria, sperm motility abnormalities are observed in these patients.
  These volunteers receive two pentoxifylline tablets(400 mg) daily for 3 month, (TRENTAL 400 mg modified release tablets, OSPS; 400 mg ,two times daily)
  Other names:
  Trental
  Interventions: Drug: Pentoxifylline
- Zinc Sulfate group (Experimental): Infertile men referred to an infertility treatment center who have had unprotected sex for at least one year have not had normal fertility in their partner. These men are all married. According to WHO criteria, sperm motility abnormalities are observed in these patients. Candidates receive one zinc sulfate tablet(229 mg) daily for 3 month,(Zinc Sulfate 220mg Capsules)
  Other Names:
  zinc sulfate
  Interventions: Drug: Zinc Sulfate 220 mg Capsules
- pentoxifylline+ zinc group (Experimental): Infertile men referred to an infertility treatment center who have had unprotected sex for at least one year have not had normal fertility in their partner. These men are all married. According to WHO criteria, sperm motility abnormalities are observed in these patients. Candidates receive one zinc sulfate(220mg) tablet+ two pentoxifylline tablets(400 mg) daily for 3 month (TRENTAL 400 mg modified release tablets, OSPS; 400 mg +Zinc Sulfate 220mg Capsules)
  Other Names:
  zinc sulfate
  Interventions: Drug: Zinc Sulfate 220 mg Capsules; Drug: Pentoxifylline

INTERVENTIONS:
Drug: Zinc Sulfate 220 mg Capsules — Zinc is an element that is involved in the activity of antioxidant enzymes. For example, the superoxide dismutase needs copper and zinc to function properly. Infertile men with asthenospermia receive 220 mg zinc sulfate tablets for 3 months
  Other Names: zinc
  Arms: Zinc Sulfate group; pentoxifylline+ zinc group
Drug: Pentoxifylline — Oral use of pentoxifylline is effective in treating cardiovascular disease, cerebrovascular disease, and other conditions associated with local circulatory disorders. Pentoxifylline affects blood viscosity. Infertile men with asthenospermia receive 400 mg pentoxifylline tablets for 3 months
  Other Names: Trental
  Arms: pentoxifylline group; pentoxifylline+ zinc group

SUMMARY:
The aim of this study was to investigate the therapeutic effect of co-administration of pentoxifylline and zinc on sperm apoptosis in men with idiopathic infertility

DETAILED DESCRIPTION:
This study is being performed as a double-blind randomized clinical trial on idiopathic infertile men referred to the infertility clinic of Shafa Clinic. Patient satisfaction, non-use of contraceptives, men aged 25 to 43 years, and idiopathic infertility according to WHO criteria (World Health, 2010) are our study criteria. Any medication that may affect the course of spermatogenesis should be discontinued during the study. Semen samples are taken from patients (before and after interventions) and apoptosis tests are performed on semen samples.

ELIGIBILITY:
Inclusion Criteria:

* infertile men
* have had at least one year of unprotected intercourse infertility
* asthenozoospermia

Exclusion Criteria:

* Men with varicocele
* Hypersensitivity to pentoxifylline & zinc,
* pelvic organic pathologies
* congenital adrenal hyperplasia
* thyroid dysfunction
* Cushing's syndrome
* hyper prolactinemia
* androgen secreting neoplasia
* severe hepatic
* pancreatitis
* kidney diseases
* gallbladder diseases
* Patients with alcohol consumption
* Patients who use cigarettes and drugs

Ages: 23 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-01-08 (Estimated); Study Completion 2022-01-20 (Estimated)

PRIMARY OUTCOMES:
sperm concentration | 1 day
  count of sperm(In per million - with the help of a neobar slide and microscopic observation
spem motility | 1 day
  motility of sperm: Calculate the percentage of motile sperm using microscopic observation
sperm morphology | 1 day
  Calculate the percentage of sperm with a normal shape with the help of Papanic staining
lipid proxidation | One week
  Malondialdehyde (nmol/mL), is measured using related experimental kits
reactive oxygen species | One week
  eactive oxygen species (ROS (RLU/s)), is measured using related experimental kits
total antioxidant capacity | One week
  total antioxidant capacity (TAC (/m / l)) is measured using related experimental kits
FSH hormon | One week
  FSH (IU / L) is measured from the blood serum of volunteers using ELISA kit
LH hormon | One week
  LH (IU / L) is measured from the blood serum of volunteers using ELISA kit
testosteron hormon [ Time Frame: One week after starting the medication ] testosterone | One week
  testosterone (nanomolar per liter) is measured from the blood serum of volunteers using ELISA kit
(Tissue necrosis Factor) | One week
  TNF α( Tissue necrosis Factor) (pg/mL) as an inflammatory factor is measured using related experimental kit
interleukin-6 | One week
  interleukin-6 (IL-6)/(pg/mL) as an inflammatory factor is measured using related experimental kit
Sperm DNA Fragmentation Assay(SDFA) | One week
  DNA fragmentation is assessed using an SDFA kit and microscopic observations (as a percentage of damaged sperm).

SECONDARY OUTCOMES:
BAX expression | 3 month
  BAX expression [ Time Frame: 3 months ]
  expression of BAX gen(in p.c) using real-time PCR and Western blot
Bcl2 expression | 3 months
  Bcl-2 gen(in p.c) using real-time PCR and Western blot
caspase 3 expression | 3 months
  expression of caspase 3 gen(in p.c) using real-time PCR and Western blot

CONTACTS AND LOCATIONS:
Overall Officials: zeynab dadgar, dr, Principal Investigator — arak university of medical science
Locations (2):
- Iran (2):
  - Infertility Center, Arak, Markazi Province
  - Arak university of medical science, Arak, Markazi Province

IPD SHARING:
Plan to Share IPD: No